CLINICAL TRIAL: NCT02521012
Title: Follow-up Study With Randomized Clinical Vitamin D Supplementation Trial on Patients With Depression (DepFuD)
Brief Title: Follow-up Study With Clinical Vitamin D Supplementation Trial on Patients With Depression (DepFuD)
Acronym: DepFuD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH5703453
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Depression; Depressive Disorder
Keywords: Depression; Depressive symptoms; Vitamin D; Intervention
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D 10 micrograms (Active Comparator): Vitamin D supplementation 10 micrograms/day given to depressed individuals, defined as "reference"
  Interventions: Dietary Supplement: Vitamin D 10 micrograms
- Vitamin D 100 micrograms (Experimental): Vitamin D supplementation 100 micrograms/day given to depressed individuals
  Interventions: Dietary Supplement: Vitamin D 100 micrograms

INTERVENTIONS:
Dietary Supplement: Vitamin D 10 micrograms — Vitamin D supplementations of 10 micrograms/day will be given to depressed individuals for three months
  Arms: Vitamin D 10 micrograms
Dietary Supplement: Vitamin D 100 micrograms — Vitamin D supplementations of 100 micrograms/day will be given to depressed individuals for three months
  Arms: Vitamin D 100 micrograms

SUMMARY:
Depression affects 350 million people worldwide. In the light of the global disease burden statistics, the efficacy of current treatments for depression appears insufficient. Thus, research on novel treatment interventions and predictors for good treatment response are warranted. Earlier prospective follow-up studies and intervention studies suggest that several bio-psychosocial factors, including high serum concentrations of vitamin D, are related to better treatment outcomes. In this follow-up study with randomized clinical vitamin D supplementation trial on patients with depression, the investigators aim to

1. clarify how a six-month intervention with vitamin D supplementation affects treatment response, recovery, and the biological pathways related to depression. This aims to finding potential sub-groups getting benefits from vitamin D supplementation. In addition, the investigators want to
2. investigate and characterize factors related to recovery from depression and working ability in depression patients in the long-term. The investigators are especially interested in the bio-psychosocial factors and the aims include examining both the individual's positive resources.

The trial will start with a six-month double-blinded randomized controlled trial with vitamin D supplementation. The aim is to recruit altogether 478 patients with non-psychotic, unipolar depression, aged 18-65 years, who are referred to the recruitment sites for treatment for depression. The participants will be randomized to low (10 µg/day) or high (100 µg/day) vitamin D supplementation group. Clinically necessary antidepressant treatments will continue during the intervention as needed. After six months of intervention, the participants will be followed up at 18 months and at 6 years.

Several measurements will be conducted during the intervention and follow-up period. Participants will fill a variety of clinical questionnaires and questionnaires with background information. All participants give blood samples for biomarker analyses at time points 3, 6, 18 months and 6 years. Clinical interviews of mental disorders (e.g. SCID) and anthropometric measurements (e.g. weight, height, blood pressure) will be carried out.

DETAILED DESCRIPTION:
Depression affects 350 million people worldwide. In the light of the global disease burden statistics, the efficacy of current treatments for depression appears insufficient. Thus, research on novel treatment interventions and predictors for good treatment response are warranted. Earlier prospective follow-up studies and intervention studies suggest that several bio-psychosocial factors, including high serum concentrations of vitamin D, are related to better treatment outcomes.

In this follow-up study with randomized clinical vitamin D supplementation trial on patients with depression, the investigators aim to

1. clarify how a six-month intervention with vitamin D supplementation affects treatment response, recovery, and the biological pathways related to depression. This aims to finding potential sub-groups getting benefits from vitamin D supplementation. In addition, the investigators want to
2. investigate and characterize factors related to recovery from depression and working ability in depression patients in the long-term. The investigators are especially interested in the bio-psychosocial factors and the aims include examining both the individual's positive resources.

The trial will start with a six-month double-blinded randomized controlled trial with vitamin D supplementation. The aim is to recruit altogether 478 patients with non-psychotic, unipolar depression, aged 18-65 years, who are referred to the recruitment sites for treatment for depression. The participants will be randomized to low (10 µg/day) or high (100 µg/day) vitamin D supplementation group. Clinically necessary antidepressant treatments will continue during the intervention as needed. After six months of intervention, the participants will be followed up at 18 months and at 6years.

Several measurements will be conducted during the intervention and follow-up period. Participants will fill a variety of clinical questionnaires and questionnaires with background information. All participants give blood samples for biomarker analyses at time points 3, 6, 18 months and 6 years. Clinical interviews of mental disorders (e.g. SCID) and anthropometric measurements (e.g. weight, height, blood pressure) will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the recruitment sites for treatment for depression
* mild, moderate or severe depression,
* mild, moderate or severe episode of recurrent depression

Exclusion Criteria:

* bipolar or psychotic depression
* psychotic disorder
* severe substance abuse
* disabilities in senses that affect functioning and severely threat completing the trial
* diseases that affect vitamin D metabolism (such as sarcoidosis, hypercalcemia, hypofunction of kidney)
* pregnancy or lactation
* current use of high dose vitamin D supplementation
* current use of high dose calcium supplementation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) scores | 0, 3 and 6 months
  We are interviewing the patients with depression with MADRS, which has been found to be a practical tool for assessing depressive symptoms in clinical trials. We are especially interest to see the change in scores during the intervention.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory (BDI) scores | 0, 3, 6, 18 months
  Participants fill a 21-item Beck Depression Inventory questionnaire and total scores will be calculated. We are especially interested to see if the total scores changes during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maarit Pakarinen, MD, PhD, Study Chair — Clinical lecturer
Locations (1):
- Welbeing Servivces County of North Savo, Kuopio University Hospital, Department of Psychiatry, Kuopio, Finland